CLINICAL TRIAL: NCT00830440
Title: A Multi-Center, Pilot Efficacy Study of the GI Sleeve™ for Pre-Surgical Weight Loss
Brief Title: A Multicenter Study for Pre-Surgical Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Morphic Medical Inc. (Industry)
Responsible Party: Principal Investigator, Jan Willem Greve, Professor, Morphic Medical Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-4
Record Dates: First submitted 2009-01-26; First posted 2009-01-28 (Estimated); Results first posted 2017-04-10 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2017-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- EndoBarrier Device (Experimental): EndoBarrier Device and Diet & Lifestyle Counseling
  Interventions: Device: EndoBarrier Device; Behavioral: Diet & Lifestyle Counseling
- Control (Active Comparator): Diet & Lifestyle Counseling
  Interventions: Behavioral: Diet & Lifestyle Counseling

INTERVENTIONS:
Device: EndoBarrier Device — NIH derived dietary, exercise and behavior modification 2005 guidelines. https://health.gov/dietaryguidelines/2005.asp and EndoBarrier Device for 12 weeks
  Other Names: EndoBarrier Gastrointestinal Liner
  Arms: EndoBarrier Device
Behavioral: Diet & Lifestyle Counseling — NIH derived dietary, exercise and behavior modification 2005 guidelines. https://health.gov/dietaryguidelines/2005.asp

SUMMARY:
The purpose of the study is to evaluate the safety and initial efficacy of the EndoBarrier device compared to a diet control in patients who require weight loss prior to their Bariatric surgery.

It is a randomized, prospective controlled, open label, pilot study of 40 patients. Thiry patients will receive an implant of the EndoBarrier device and the other 10 patients will receive the principle investigator's standard of care diet program. All patients will be treated for 12 weeks with the exception of the last 10 device patients who will continue to 24 weeks if the principle investigator determines that it is safe and in their best interest to continue.

The primary efficacy endpoint is:

* Assessment of the difference in % excess weight loss between the 2 groups

Secondary endpoints are:

* Resolution or Improvement in type II Diabetic status as defined as:
* Resolution = patient is off their diabetes medication and has normal diabetic blood parameters (fasting glucose)
* Improvement = normalizing diabetic blood parameters (fasting glucose) and/or a reduction in dosing or frequency of their diabetic medication
* The percent of patients who achieve at least a 10% excess weight loss will be calculated as a secondary outcome.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years and < 55 years - Male or Female
* BMI > 35 with significant comorbidities (i.e. hypertension, or hyperlipidemia, or diabetes) or > 40 BMI <60 (with or without a co-morbid condition)
* History of failure with nonsurgical weight loss methods
* Candidates for Roux-en-Y gastric bypass
* Patients willing to comply with study requirements
* Patients who have signed an informed consent form

Exclusion Criteria:

* Patients requiring prescription anticoagulation therapy
* Patients with iron deficiency and iron deficiency anemia
* Inflammatory bowel disease or condition of the gastrointestinal tract, such as ulcers or Crohn's disease
* Treatment represents an unreasonable risk to the patient
* Pancreatitis or other serious organic conditions
* Symptomatic coronary artery disease or pulmonary dysfunction
* Patients with known gallstones prior to implant
* Known infection at the time of implant
* Severe coagulopathy, upper gastro-intestinal bleeding conditions such as esophageal or gastric varices, congenital or acquired intestinal telangiectasia
* Congenital or acquired anomalies of the GI tract such as atresias or stenoses
* Pregnant or has the intention of becoming pregnant in the next 12 months
* Unresolved alcohol or drug addiction
* HIV Positive patients
* Patients with hepatitis B or C
* Mentally retarded or emotionally unstable, or exhibits psychological characteristics which, in the opinion of the investigator, makes the subject a poor candidate for device placement or clinical trial
* Previous GI surgery that could affect the ability to place the sleeve or the function of the implant.
* Patients unable to discontinue NSAIDs (non-steroidal anti-inflammatory drugs) during the implant period
* H. pylori positive patients (Note: patients may be enrolled if they had a prior history and were successfully treated)
* Patients receiving weight loss medications such as Meridia and Xenical
* Family or patient history of a known diagnosis or pre-existing symptoms of systemic lupus erythematosus, scleroderma or other autoimmune connective tissue disorder
* Patients with gastroesophageal reflux disease (GERD)
* Patients with a history of kidney stones
* Participating in another ongoing investigational clinical trial

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2007-01; Primary Completion 2008-03 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Willem Greve, MD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- University Hospital Maastricht, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schouten R, Rijs CS, Bouvy ND, Hameeteman W, Koek GH, Janssen IM, Greve JW. A multicenter, randomized efficacy study of the EndoBarrier Gastrointestinal Liner for presurgical weight loss prior to bariatric surgery. Ann Surg. 2010 Feb;251(2):236-43. doi: 10.1097/SLA.0b013e3181bdfbff. PMID 19858703

RESULTS

PARTICIPANT FLOW:
Groups:
- EndoBarrier Device: EndoBarrier + Diet + Lifestyle counseling 12 Week implant duration
  EndoBarrier: Monthly visits
- Control (Diet & Lifestyle Counseling): Diet + Lifestyle counseling
  Diet + Lifestyle Counseling: Monthly Visits
Period: Overall Study
Arm/Group | EndoBarrier Device | Control (Diet & Lifestyle Counseling)
Started | 32 | 11
Received Device | 26 | 0
Completed 12 Week Follow up | 24 | 11
Completed 16 Week Follow up | 4 | 0
Completed 24 Week Follow up | 3 | 0
Completed | 24 | 11
Not Completed | 8 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — unsuccessful procedure | 4 | 0
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Population: EndoBarrier subjects with a successful implant
Groups:
- EndoBarrier and Diet/Lifestyle Counseling: EndoBarrier + Diet + Lifestyle counseling
  EndoBarrier: Monthly visits
- Control: (Diet and Lifestyle Counseling): Diet + Lifestyle counseling
  Diet + Lifestyle Counseling: Monthly Visits
- Total: Total of all reporting groups
Arm/Group | EndoBarrier and Diet/Lifestyle Counseling | Control: (Diet and Lifestyle Counseling) | Total
Number analyzed (Participants) | 26 | 11 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.9 (9.33) | 41.2 (10.46) | 41.0 (9.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 9 | 27
  Male | 8 | 2 | 10
Region of Enrollment [Number; unit: participants]
  Netherlands | 26 | 11 | 37

OUTCOME MEASURES:

1. Primary Outcome: Total Weight Change From Baseline at 12 Weeks in kg
Time Frame: 12 weeks
Population: 26 subjects received the device. 2 subjects had the device removed before 12 weeks.
Measure: Mean (Standard Deviation); unit: kg
Groups:
- EndoBarrier/Diet and Lifestyle Counseling/12 Weeks: 12 week implantation period
Arm/Group | EndoBarrier/Diet and Lifestyle Counseling/12 Weeks | Control (Diet & Lifestyle Counseling)
Number analyzed (Participants) | 24 | 11
kg | -13.3 (5.83) | -5.5 (5.41)

2. Secondary Outcome: % of Subjects Achieving at Least a 10% Change in Excess Weight From Baseline to 12 Weeks
Description: The percent excess weight loss calculated using the Metropolitan Life Tables (MET). The actual amount of excess weight loss (EWL) was examined through the percent of actual weight change from baseline.
Time Frame: 12 weeks
Measure: Number; unit: % participants
Groups:
- EndoBarrier and Diet and Lifestyle Counseling: EndoBarrier + Diet + Lifestyle counseling
  EndoBarrier: Monthly visits
Arm/Group | EndoBarrier and Diet and Lifestyle Counseling | Control (Diet & Lifestyle Counseling)
Number analyzed (Participants) | 24 | 11
% participants | 80.8 | 27.3

3. Secondary Outcome: Count of Subjects With Decrease in HbA1c Values From Baseline to Week 12
Time Frame: Baseline to Week 12 of treatment
Population: Type 2 Diabetes Subjects
Measure: Count of Participants; unit: Participants
Arm/Group | EndoBarrier/Diet and Lifestyle Counseling/12 Weeks | Control (Diet & Lifestyle Counseling)
Number analyzed (Participants) | 8 | 2
Participants | 8 | 1

ADVERSE EVENTS:
Arm/Group | EndoBarrier and Diet and Lifestyle Counseling | Control (Diet & Lifestyle Counseling)
Serious Adverse Events (participants affected / at risk) | 1/26 | 0/11
Other Adverse Events (participants affected / at risk) | 26/26 | 1/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EndoBarrier and Diet and Lifestyle Counseling (N=26) | Control (Diet & Lifestyle Counseling) (N=11)
Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EndoBarrier and Diet and Lifestyle Counseling (N=26) | Control (Diet & Lifestyle Counseling) (N=11)
Abdominal pain upper (Gastrointestinal disorders) | 13 (20) | 0 (0)
Adverse drug reaction (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 8 (8) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 7 (7) | 0 (0)
Implant site inflammation (Injury, poisoning and procedural complications) | 5 (5) | 0 (0)
Nausea (Gastrointestinal disorders) | 11 (12) | 1 (1)
Polyp (Gastrointestinal disorders) | 2 (2) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 9 (9) | 0 (0)
Procedural vomiting (Gastrointestinal disorders) | 4 (4) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No